CLINICAL TRIAL: NCT02968927
Title: A Ph2 Randomized Trial to Evaluate the Safety Preliminary Efficacy and Biomarker Response of Host Directed Therapies Added to Rifabutin-modified Standard Therapy in Adults With Drug-Sensitive Smear-Positive Pulmonary TB
Brief Title: TB Host Directed Therapy
Acronym: TBHDT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Aurum Institute NPC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TBHDT-AUR1-8-178
Record Dates: First submitted 2016-09-08; First posted 2016-11-21 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Everolimus; Auranofin; Cholecalciferol; CC-11050

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 2HRbEZ/4HRb (Active Comparator): 2HRbZE
  Interventions: Drug: 2HRbZE/4HRb
- Everolimus (Experimental): Everolimus 0.5 MG
  Interventions: Drug: Everolimus 0.5 MG; Drug: 2HRbZE/4HRb
- Auranofin (Experimental): Auranofin 6 MG
  Interventions: Drug: Auranofin 6 MG; Drug: 2HRbZE/4HRb
- Vitamin D (Experimental): Vitamin D3
  Interventions: Drug: Vitamin D3; Drug: 2HRbZE/4HRb
- CC-11050 (Experimental): CC-11050
  Interventions: Drug: CC-11050; Drug: 2HRbZE/4HRb

INTERVENTIONS:
Drug: Everolimus 0.5 MG
  Arms: Everolimus
Drug: Auranofin 6 MG
  Arms: Auranofin
Drug: Vitamin D3
  Arms: Vitamin D
Drug: CC-11050
  Arms: CC-11050
Drug: 2HRbZE/4HRb
  Other Names: rifabutin-modified TB therapy

SUMMARY:
To examine the safety and preliminary efficacy of multiple adjunctive host directed TB therapies (TB HDT), to assess their potential to shorten TB treatment and/or prevent permanent lung damage.

DETAILED DESCRIPTION:
OBJECTIVES:

To determine the safety and preliminary efficacy of 4 TB HDT candidates:

1. Safety (treatment emergent serious adverse events and SUSARs)
2. Microbiologic effects in sputum (culture conversion, change in MGIT TTP) and blood (WBA)
3. PET/CT imaging
4. Serum markers of inflammation
5. Effects on Mtb-specific and general immune function
6. Pulmonary effects (spirometry, 6MWT, O2 saturation, and St. George Respiratory Symptom Questionnaire) In each case, TB HDT effects will be determined by comparison to patients treated with standard TB therapy alone with regard to a common set of primary and secondary endpoints.

PRIMARY ENDPOINTS

1. For auranofin, everolimus, and vitamin D: the proportions of patients experiencing suspected unexpected serious adverse reactions (SUSARs).
2. For CC-11050: the proportion of patients experiencing treatment emergent serious adverse events (SAEs).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide signed written consent or witnessed oral consent in the case of illiteracy, prior to undertaking any trial-related procedures.
2. Aged 18 to 65 years, male, or if female, either not of reproductive potential (post-menopause, or status-post surgical sterilization) or with an intrauterine contraceptive device in place.
3. Body weight (in light clothing without shoes) between 40 and 90 kg.
4. First episode of pulmonary tuberculosis diagnosed by positive sputum AFB smear with subsequent culture confirmation OR positive Xpert TB/RIF with Ct <20 [4].
5. RIF susceptibility diagnosed by Xpert TB/RIF OR Hain test
6. Chest radiograph meeting criteria for moderate or far advanced pulmonary tuberculosis [5]
7. HIV-1 seronegative
8. HBsAg negative

Exclusion Criteria:

1. Any condition for which participation in the trial, as judged by the investigator, could compromise the well-being of the subject or prevent, limit or confound protocol specified assessments
2. Current or imminent treatment for malaria.
3. Is critically ill, and in the judgment of the investigator has a diagnosis likely to result in death during the trial or the follow-up period.
4. TB meningitis or other forms of severe tuberculosis with high risk of a poor outcome as judged by the investigator.
5. History of allergy or hypersensitivity to any of the trial therapies or related substances, including known allergy or suspected hypersensitivity to rifampin or rifabutin.
6. Having participated in other clinical trials with investigational agents within 8 weeks prior to trial start or currently enrolled in an investigational trial.
7. Subjects with any of the following at screening:

   1. Cardiac arrhythmia requiring medication;
   2. Prolongation of QT/QTc interval with QTcF (Fridericia correction) >450 ms;
   3. History of additional risk factors for Torsade de Pointes, (e.g., heart failure, hypokalemia, family history of Long QT Syndrome);
   4. Any clinically significant ECG abnormality, in the opinion of the investigator.
   5. Patients requiring concomitant medications that prolong the QT inter-val.
8. Random blood glucose >140 mg/dL, or history of unstable Diabetes Mellitus which required hospitalization for hyper- or hypoglycaemia within the past year prior to start of screening.
9. Use of systemic corticosteroids within the past 28 days.
10. Subjects with any of the following abnormal laboratory values:

    1. creatinine >2 mg/dL
    2. haemoglobin <8 g/dL
    3. platelets <100x109 cells/L
    4. serum potassium <3.5
    5. aspartate aminotransferase (AST) ≥2.0 x ULN
    6. alkaline phosphatase (AP) >5.0 x ULN
    7. total bilirubin >1.5 mg/dL

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
SAEs and SUSARs | through day 180
  For auranofin, everolimus, and vitamin D: the proportions of patients experiencing suspected unexpected serious adverse reactions (SUSARs).
  For CC-11050: the proportion of patients experiencing treatment emergent serious adverse events (SAEs).

SECONDARY OUTCOMES:
TEAEs other than SAEs and SUSARs | through day 180
  TEAEs other than SAEs, categorized according to severity, drug relatedness, and leading to early withdrawal.
Sputum culture status on day 56 | day 56
  Proportion of patients with positive sputum cultures on solid culture medium after 8 weeks of treatment

OTHER OUTCOMES:
Change in FEV1 from baseline to 2 and 6 months | days 56 and 180
  FEV1 (% of expected value)
18F-FDG PET/CT imaging (change from baseline to 2 months): | day 56
  Maximum and mean standardized uptake values (SUV)
Serum neopterin | day 56
  change from baseline b. CRP
Quantiferon gold in tube | day 56
  change from baseline
Gene expression profiles (exploratory) | days 56 and 180
  Change from baseline to 2 and 6 months in gene expression profiles
PD-1 expression (exploratory) | days 56 and 180
  PD-1 expression on CD4 and CD8 lymphocytes

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Wallis, MD,FIDSA, Principal Investigator — The Aurum Institute NPC
Locations (1):
- The Aurum Institute: Tembisa Clinical Research Centre, Tembisa, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wallis RS, Ginindza S, Beattie T, Arjun N, Likoti M, Edward VA, Rassool M, Ahmed K, Fielding K, Ahidjo BA, Vangu MDT, Churchyard G. Adjunctive host-directed therapies for pulmonary tuberculosis: a prospective, open-label, phase 2, randomised controlled trial. Lancet Respir Med. 2021 Aug;9(8):897-908. doi: 10.1016/S2213-2600(20)30448-3. Epub 2021 Mar 16. PMID 33740465